CLINICAL TRIAL: NCT06078735
Title: Vascular Closure With Novel Ergonomic External Compression Device Compared to Manual Compression After Atrial Fibrillation Ablation: The LockeT II Study
Brief Title: Vascular Closure With a Device Compared to Manual Compression After Atrial Fibrillation Ablation: The LockeT II Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KCHRRF_LockeT II_0023
Record Dates: First submitted 2023-09-21; First posted 2023-10-12 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation; Hemostasis
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to LockeT device or Manual Compression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LockeT (Experimental): These are the patients assigned for LockeT device arm to close the access site wound.
  Interventions: Device: Vascular closure with LockeT device
- Manual compression (No Intervention): These are the patients assigned for Manual Compression arm to close the access site wound.

INTERVENTIONS:
Device: Vascular closure with LockeT device — For subjects that are assigned to the LockeT device arm, the healthcare professional will place the LockeT with suture above the wound to achieve compression instead of manually holding pressure on the sutures. After hemostasis is achieved and prior to ambulation the LockeT will be removed followed by suture removal.
  Arms: LockeT

SUMMARY:
The LockeT II study is a single center, prospective randomized study. It is intended to study the effectiveness of using LockeT device to gain hemostasis after venous procedures as compared to Manual Compression (MC). Approximately 110 patients will be enrolled.

DETAILED DESCRIPTION:
The volume of catheter ablation procedures for the treatment of atrial fibrillation and other arrhythmias are on the rise in the United States and worldwide. Despite decrease in complication rates due to refinement in ablation tools and techniques, achieving vascular hemostasis following large-bore sheath femoral access remains a challenge. Thus, MC remains the current standard of care. However, MC requires up to 8 hours of prolonged bedrest, which is associated with longer length of stay and complications from indwelling catheters.

Another method of vascular closure is the figure-of-eight (FoE) stitch - a subcutaneous suture that has been evaluated to achieve homeostasis following major cardiovascular procedures.

In recent years, invasive, vascular closure devices have become popular. However, results continue to suggest that the risk versus benefit has not been definitively demonstrated. Instead, the LockeT is a new suture retention device designed to closely mimic manual compression by distributing the tension of a FoE stitch over a larger surface area. In such a way, patients can have the benefits of MC without a healthcare professional to stand bedside.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Be able to provide consent
* Presenting for planned procedures that require percutaneous venous punctures, such as atrial fibrillation radiofrequency ablation, and where the physician utilizes a LockeT device or MC to close the wound.

Exclusion Criteria:

* Under the age of 18
* Unable to or unwilling to provide consent
* Cannot comply with study requirements
* Not undergoing procedures that require a percutaneous venous puncture or planned access to the left atrium and/or ventricle
* Subjects whose physician does not use LockeT or MC to close the venous puncture.
* Patient is currently pregnant, as evidenced by positive urine Beta-HCG. (Urine Beta Human chorionic gonadotropin (HCG) will be checked in all females of the reproductive age group).
* If the physician detects a formed hematoma prior to venous closure, that patient will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of using the LockeT suture retention device | 2 Days
  Effectiveness of using the LockeT suture retention device to gain hemostasis after venous procedures as compared to standard Manual Compression (MC) will be assessed.

SECONDARY OUTCOMES:
Patient, physician, and nursing staff benefits | 2 Days
  Patient, physician, and nursing staff benefits of the LockeT device will be assessed via LockeT device questionnaire with a scale of 1 to 5, 1 strongly disagree and 5 strongly agree.
Patient discomfort with Locket device | 2 Days
  Pain discomfort will be assessed via Locket device questionnaire with a scale of 1 to 5, 1 strongly disagree and 5 strongly agree.
Incidence of hematoma/ecchymosis | 2 Days
  The incidence of hematoma/ecchymosis post-procedure will be assessed.
Safety of LockeT device | 2 Days
  Safety of LockeT device will be assessed by the incidence of adverse events, including but not limited to: vascular complications, like atrioventricular (AV) fistula, retroperitoneal bleed, surgical exploration of the groin (thrombin injection, open surgery or ligation); need for blood transfusion, defined as a 2 gm post-procedure drop in hemoglobin, or symptoms of anemia,).
Comparison of Manual Compression labor cost and Locket device cost | 2 Days
  Manual Compression labor cost and Locket device cost will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (6):
- United States (6):
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center Clinic, Independence, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

REFERENCES:
- [Background] Natale A, Mohanty S, Liu PY, Mittal S, Al-Ahmad A, De Lurgio DB, Horton R, Spear W, Bailey S, Bunch J, Musat D, O'Neill P, Compton S, Turakhia MP; AMBULATE Trial Investigators. Venous Vascular Closure System Versus Manual Compression Following Multiple Access Electrophysiology Procedures: The AMBULATE Trial. JACC Clin Electrophysiol. 2020 Jan;6(1):111-124. doi: 10.1016/j.jacep.2019.08.013. Epub 2019 Oct 30. PMID 31971899
- [Background] Mujer MT, Al-Abcha A, Flores J, Saleh Y, Robinson P. A comparison of figure-of-8-suture versus manual compression for venous access closure after cardiac procedures: An updated meta-analysis. Pacing Clin Electrophysiol. 2020 Aug;43(8):856-865. doi: 10.1111/pace.14008. Epub 2020 Jul 20. PMID 32638389
- [Background] Atti V, Turagam MK, Garg J, Alratroot A, Abela GS, Rayamajhi S, Lakkireddy D. Efficacy and safety of figure-of-eight suture versus manual pressure for venous access closure: a systematic review and meta-analysis. J Interv Card Electrophysiol. 2020 Apr;57(3):379-385. doi: 10.1007/s10840-019-00547-6. Epub 2019 Apr 18. PMID 31001767
- [Background] Jensen CJ, Schnur M, Lask S, Attanasio P, Gotzmann M, Kara K, Hanefeld C, Mugge A, Wutzler A. Feasibility of the Figure-of-8-Suture as Venous Closure in Interventional Electrophysiology: One Strategy for All? Int J Med Sci. 2020 Apr 6;17(7):965-969. doi: 10.7150/ijms.42593. eCollection 2020. PMID 32308550